CLINICAL TRIAL: NCT03185416
Title: Early Palliative Care Integration in Interventional Cancer Care
Acronym: EPIICC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving University
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ana M. Echenique, Associate Professor of Clinical, Vascular Interventional, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20161049
Record Dates: First submitted 2017-04-27; First posted 2017-06-14 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Palliative Care; Cancer Liver; Cancer Colon
Keywords: Quality of Life; Caregiver; Quality Improvement
MeSH Terms: conditions — Carcinoma, Hepatocellular; Colonic Neoplasms | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: The present study is a randomized single-center therapeutic clinical trial including the following two prospective groups: Control group and the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The first prospective group -the control group- will consist of 30 patients receiving treatment by the Interventional Radiology team- along with their 30 primary caregivers. Neither the patient nor the caregiver will receive the palliative care training intervention. Patients and their caregivers will receive questionnaires regarding their health status (physical and psychosocial) and health services utilization at 1, 2, and 3 months post-procedure- during their follow-up visits.
- Intervention Group (Experimental): The second prospective component of the study -the intervention group- will include 30 patients receiving treatment by the Interventional Radiology team along with their primary caregiver. Patients and caregivers will receive a brief palliative care training intervention during their first follow-up visit. Patients and their caregivers will receive questionnaires to assess their health status (physical and psychosocial) and health services utilization outcomes at 1, 2, and 3 months post-procedure during their follow-up visits.
  Interventions: Other: Palliative Care Training

INTERVENTIONS:
Other: Palliative Care Training — The intervention group- will include 30 patients receiving treatment by the Interventional Radiology team along with their primary caregiver. Patients and caregivers will receive a brief palliative care training intervention during their first follow-up visit. Patients and their caregivers will receive questionnaires to assess their health status (physical and psychosocial) and health services utilization outcomes at 1, 2, and 3 months post-procedure during their follow-up visits.
  Other Names: Counseling
  Arms: Intervention Group

SUMMARY:
A mixed methods randomized control trial assessing the impact of early palliative care incorporation in liver cancer and metastatic colorectal cancer on caregiver well-being, patient physical and psychosocial outcomes, and health services utilization.

DETAILED DESCRIPTION:
The purpose of this project is to conduct a mixed-methods study of the impact of early integration of palliative care in interventional oncology on three outcomes of interest:

1) caregiver well-being, 2) patient physical and psychosocial outcomes, and 3) health services utilization and costs. Palliative care focuses on providing patients with serious illnesses and their families with physical, emotional, social, practical, and spiritual support. Recent trials examining the integration of palliative care in cancer care have individually shown improvement in patient symptoms and quality of life, reduction of caregiver burden, and/or health services costs. These studies, however, have not collectively analyzed these impacts.Further, a recent study shows that integrating palliative care early in lung cancer care has proven beneficial to both patients and caregivers. Given the potential of this previous body of research, the proposed study offers a comprehensive analysis of the early integration of palliative care on caregiver well-being, patient's physical and psychosocial outcomes when living with liver and metastatic colorectal cancer (mCRC), and health services utilization. This study thus broadens the scope to additional cancer types and degrees of progression.

ELIGIBILITY:
Inclusion Criteria:

- Patients over 18 years of age with a confirmed diagnosis of liver cancer or metastatic colorectal cancer requiring treatment from the IR team.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Edmonton Symptom Assessment Score (ESAS-R) | 1, 2 and 3 months
  Measure the impact of an early palliative care intervention on patient physical and psychosocial outcomes. The early integration of palliative care at diagnosis or immediately post- procedure, will improve patients' physical and psychosocial symptoms. The score of such assessment should decrease from baseline as the result of the intervention.

SECONDARY OUTCOMES:
Measure of the Eastern Cooperative Oncology Group (ECOG) performance Status | 1, 2 and 3 months
  Measure the decrease of the ECOG status as a result of the proposed intervention.

OTHER OUTCOMES:
Caregiver Well-being Scale | 1, 2 and 3 months
  The caregiver well-being Scale will measure the Caregiver Well-Being.
Caregiver Quality of Life-Cancer Scale | 1, 2 and 3 months
  The caregiver Quality of Life-Cancer Scale will measure the quality of life of subjects with cancer.
Measure the decrease in the score of the Center for Epidemiologic Studies Depression Scale (CES-D). | 1, 2 and 3 months
  It is anticipated that the CES-D score will be decreased from baseline as a result of the proposed intervention.
Health services utilization | 1, 2 and 3 months
  Subsequent to the integration of palliative care resulting in improved patient outcomes, the frequency of ED visits, ICU visits, and hospital stays will decrease.
Health services costs | 1, 2 and 3 months
  Subsequent to the integration of palliative care resulting in improved patient outcomes, the frequency of ED visits, ICU visits, and hospital stays will decrease and therefore reduce costs.

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Echenique, MD, Principal Investigator — Univeristy of Miami

IPD SHARING:
Plan to Share IPD: Undecided
There are no plans to share IPD with other researchers.